CLINICAL TRIAL: NCT02575131
Title: The Effect of Breakfast Test Products on Acute Satiety Scores in Different Test Conditions
Brief Title: Breakfast Test Products and Acute Satiety Scores
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Nederlands Bakkerij Centrum (Other); PepsiCo, Inc. (Industry)
Responsible Party: Principal Investigator, W.J. Pasman, Consultant Clinical Trials, TNO
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 9619
Record Dates: First submitted 2015-10-06; First posted 2015-10-14 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
Keywords: satiety; overweight; breakfast; ecological validity
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- TNO whole wheat bread yeast basis (Experimental): NBC-1: four slices of whole wheat bread yeast basis (98 grams) spread with 3 cups low-fat margarine (total 30 grams) consumed with 200 mL of black coffee (without milk and sugar) or 200 mL tea (no sugar) or 200 mL of water at TNO
  Interventions: Other: whole wheat bread yeast basis
- TNO whole wheat sourdough bread (Active Comparator): NBC-2- four slices of whole wheat sourdough bread (98 grams) with 3 cups low-fat margarine (total 30 grams) consumed with 200 mL of black coffee (without milk and sugar) or 200 mL tea (no sugar) or 200 mL of water. at TNO
  Interventions: Other: whole wheat sourdough bread
- TNO Oatmeal (Experimental): PepsiCo, Inc.-1 - One portion of Steel Cut oatmeal: 66.8 grams of oats boiled for 25 minutes in 500 grams of water and consumed with 307 grams of skimmed milk at TNO
  Interventions: Other: Oatmeal
- TNO original Cheerios (Active Comparator): PepsiCo, Inc.-2 - One portion of original Cheerios (ready to eat cereal): 70 grams prepared with 307 grams of skimmed milk and consumed with about 275 grams of water at TNO
  Interventions: Other: Cheerios
- TNO standard breakfast (Experimental): TNO breakfast: one slice of white bread with a fried egg and 200 mL orange juice. With spray oil a frying pan is prepared to fry an egg (medium size).
  The breakfast is consumed at TNO
  Interventions: Other: standard breakfast
- Home whole wheat bread yeast basis (Experimental): NBC-1: four slices of whole wheat bread yeast basis (98 grams) spread with 3 cups low-fat margarine (total 30 grams) consumed with 200 mL of black coffee (without milk and sugar) or 200 mL tea (no sugar) or 200 mL of water at home
  Interventions: Other: whole wheat bread yeast basis
- Home whole wheat sourdough bread (Active Comparator): NBC-2- four slices of whole wheat sourdough bread (98 grams) with 3 cups low-fat margarine (total 30 grams) consumed with 200 mL of black coffee (without milk and sugar) or 200 mL tea (no sugar) or 200 mL of water at home
  Interventions: Other: whole wheat sourdough bread
- Home Oatmeal (Experimental): PepsiCo, Inc.-1 - One portion of Steel Cut oatmeal: 66.8 grams of oats boiled for 25 minutes in 500 grams* of water and consumed with 307 grams of skimmed milk at home
  Interventions: Other: Oatmeal
- Home original Cheerios (Active Comparator): PepsiCo, Inc.-2 - One portion of original Cheerios (ready to eat cereal): 70 grams prepared with 307 grams of skimmed milk and consumed with about 275 grams of water at home
  Interventions: Other: Cheerios
- Home standard breakfast (Experimental): one slice of white bread with a fried egg and 200 mL orange juice. With spray oil a frying pan is prepared to fry an egg (medium size).
  The breakfast is consumed at home
  Interventions: Other: standard breakfast

INTERVENTIONS:
Other: whole wheat bread yeast basis
  Arms: Home whole wheat bread yeast basis; TNO whole wheat bread yeast basis
Other: Oatmeal
  Arms: Home Oatmeal; TNO Oatmeal
Other: Cheerios
  Arms: Home original Cheerios; TNO original Cheerios
Other: whole wheat sourdough bread
  Arms: Home whole wheat sourdough bread; TNO whole wheat sourdough bread
Other: standard breakfast
  Arms: Home standard breakfast; TNO standard breakfast

SUMMARY:
Rationale: The worldwide prevalence of obesity increases rapidly, and at the moment there are more overweight than underweight people in the world. This is partly caused by increased energy, or food intake. One of the physiological factors regulating the food intake pattern is satiety. Though the regulation of food intake has been studied quite extensively, the underlying mechanisms are not well elucidated yet and still new factors involved in this regulation are being found. Therefore, in this study the investigators aim to develop an in vitro screening tool combined with an in silico model for prediction of satiety, for cost- and time - effective screening of satiating properties of new and existing complex food products and (functional) ingredients, based on actual satiety scores measured. A second aim of the Wholegrain Satiety project is to evaluate satiating properties of different types of wholegrain breads and other oat based products, both for validation purposes and to strengthen the scientific evidence for health benefits of wholegrain products. As part of this study, acute satiety scores after consumption of various breakfast products in well-controlled clinical conditions will be compared with satiety scores obtained in 'at home' test conditions.

Objective: The current study aims to compare the acute satiety effect of carbohydrate breakfast products.

DETAILED DESCRIPTION:
In the present study the investigators will conduct a clinical trial in which a standard protocol will be used to examine five different breakfasts (different in type: breakfast cereals and bread, and macronutrient composition) with satiating ingredients which will reveal actual human satiety scores. The visual analogue scales used for determination of satiety feelings is an accepted method by EFSA and studied extensively. It is used by TNO in an earlier carbohydrate containing breakfast experiment.

Subjects may feel and eat differently at home. Especially since supervision by a researcher is known to influence behavior of participants. Self-measuring has the potential of giving more reliable estimates of intervention effects. Therefore, it is interesting to repeat the tests that are performed in the clinical unit, in an 'at home' condition, because that is the place consumers eat their breakfast habitually (= ecological validity).

Study design: The study is designed as an open, randomized, controlled, cross-over trial.

Study population: Forty healthy, lean and overweight, non-restrained eating women.

Intervention: The intervention consists of five different normal breakfasts (normal amount, about 243-355 kCal; bread, cooked oatmeal, cereal meal, fried egg with bread) provided as a breakfast in the metabolic ward and at home.

Main study parameters/endpoints: Satiety scores will be obtained with visual analogue rating scales (VAS). Subjects will rate hunger feelings, fullness feelings, satiety feelings, desire to eat and rate their prospective food consumption, before and multiple times after consumption of a breakfast. A test session lasts for four hours (t = 0, 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 minutes).

In the controlled conditions at TNO, finger pricks will be performed at t = 0, 30, 60, 90 and 120 minutes after breakfast consumption to measure blood glucose.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects will consume prescribed, standardized breakfast products; five times at a clinical unit and five times at home. No risk is associated with intake of the test products. The VAS questionnaire will be filled in on the laptop multiple times on all test days (at home and at the clinic). No risk or real burden is of concern in this study. Subjects will perform finger pricks five times in each controlled session at TNO, what is known as a minimally invasive technique to obtain drops of blood.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged 18-50 years;
2. BMI: 22-32 kg/m2;
3. Written consent regarding participation after full information regarding all details of the study;
4. Normal Dutch eating habits (consuming mostly three main meals per day; used to eat bread for lunch; used to consume dietary fibres; like the test products (P9619 F02));
5. Normal dietary eating behaviour (non-restrained eaters, estimated with the Dutch Eating Behaviour Questionnaire; P9619 F06);
6. Healthy as assessed by the Health and Lifestyle questionnaire (P9619 F02);
7. Subjects with a normal dietary fibre intake (between 10-30 grams/day) (P9619 F07);
8. Voluntary participation;
9. Willing to comply with study procedures;
10. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data by TNO;
11. Have a laptop with adequate internet access at home and experience how to use it, and willing to use and bring it to TNO.

Exclusion Criteria:

1. On-going or recent treatment for diabetes, hypertension, coronary heart disease, psychiatric conditions, inflammatory chronic disease - rheumatoid arthritis, Crohn Disease, ulcerous colitis, chronic constipation, eating disorders;
2. Reported postmenopausal;
3. Having menstruation problems, e.g. PCOS;
4. Reported to be on a slimming diet or other dietary treatment (currently or during last two months, like vegetarian diet, lactose restricted diet etc.);
5. On-going use of any slimming preparations;
6. Any kind of dysfunction of digestive tract, food allergies/intolerances related to the supplied test products (like gluten intolerance), chronic constipation, recent/actual gastroenteritis;
7. Reported unexplained weight loss or gain of > 2 kg in the three months prior to the pre-study screening
8. Smoking;
9. Subjects with a high level of physical activity (> 5h intense sporting activity/week);
10. Heavy alcohol consumers, no more than 14 units per week (1 unit represents 1 standard glass/portion of alcohol, independent of the type of alcoholic drink);
11. Physical, mental or practical limitations in using computerized systems;
12. Partner or first or second-degree relative from TNO personnel stationed at TNO Zeist.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Hunger and satiety feelings for different compositions of breakfasts | four hours
  Response in hunger and satiety feelings due to breakfast consumption over time (four hours) will be measured with a visual analogue rating scale varying of no hunger (0 mm) to very hungry (100 mm)

SECONDARY OUTCOMES:
Level of control of the conduct (controlled at TNO versus less control at home) | Four hour follow-up on hunger and satiety feelings after each breakfast session
  The differences in hunger and satiety scores measured with visual analogue rating scales will be monitored for four hours after breakfast consumption at TNO (controlled setting) versus at home (less control)
Blood glucose | two hours
  In the controlled condition at TNO the blood glucose response will be monitored with finger pricks and direct blood glucose measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Wilrike J Pasman, PhD, Principal Investigator — TNO
Locations (1):
- TNO Quality of Life, Zeist, Utrecht, Netherlands

REFERENCES:
- [Background] Blundell J, de Graaf C, Hulshof T, Jebb S, Livingstone B, Lluch A, Mela D, Salah S, Schuring E, van der Knaap H, Westerterp M. Appetite control: methodological aspects of the evaluation of foods. Obes Rev. 2010 Mar;11(3):251-70. doi: 10.1111/j.1467-789X.2010.00714.x. Epub 2010 Jan 29. PMID 20122136
- [Result] Raben A, Tagliabue A, Astrup A. The reproducibility of subjective appetite scores. Br J Nutr. 1995 Apr;73(4):517-30. doi: 10.1079/bjn19950056. PMID 7794869
- [Result] Pasman WJ, Blokdijk VM, Bertina FM, Hopman WP, Hendriks HF. Effect of two breakfasts, different in carbohydrate composition, on hunger and satiety and mood in healthy men. Int J Obes Relat Metab Disord. 2003 Jun;27(6):663-8. doi: 10.1038/sj.ijo.0802284. PMID 12833109
- [Result] Marschollek M, Gietzelt M, Schulze M, Kohlmann M, Song B, Wolf KH. Wearable sensors in healthcare and sensor-enhanced health information systems: all our tomorrows? Healthc Inform Res. 2012 Jun;18(2):97-104. doi: 10.4258/hir.2012.18.2.97. Epub 2012 Jun 30. PMID 22844645
- See also: Prevalence of obesity — http://www.who.int/mediacentre/factsheets/fs311/en/#